CLINICAL TRIAL: NCT00165269
Title: Mantle Irradiation for Selected Hodgkin's Disease Patients With Stage IA-IIA Disease
Brief Title: Mantle Irradiation for Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Peter Mauch, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 92-035
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Hodgkin's Disease
Keywords: Hodgkin's Disease Stage IA-IIA; mantle irradiation
MeSH Terms: conditions — Hodgkin Disease

INTERVENTIONS:
Procedure: Mantle irradiation — Limited to above the diaphragm

SUMMARY:
The purpose of this study it to evaluate the effectiveness of radiation therapy limited to above the diaphragm in patients with pathological stage IA-IIA Hodgkin's disease.

DETAILED DESCRIPTION:
* Eligble patients will receive a course of radiation therapy directed to above the diaphragm only.
* Patients would have bloodwork and chest x-rays performed 4 times per year for the first two years, 3 times per year for the third year, and 2 times per year for the fourth and fifth years. After five years, yearly check-ups are performed.
* In addition to the above follow-up, patients will receive, once or twice a year for the first 5 years, an abdominal-pelvic CT scan and/or gallium scan.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically Stage IA-IIA Hodgkin's disease
* A negative staging laparotomy including splenectomy, biopsies of liver, paraortic nodal biopsies and palpitation of upper pelvic nodes
* 18 years of age or older

Exclusion Criteria:

* Patients with large mediastinal adenopathy
* Patients with LD histology
* Patients with "B" symptoms
* Positive laparotomy
* Subcarinal, hilar, or cardiac lymph node involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1992-05; Primary Completion 2000-06 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the risks and benefits of mantle field irradiation alone in treating Hodgkin disease patients. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mauch, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts